CLINICAL TRIAL: NCT04121897
Title: TEMPO: A Feasibility Study of a Therapist-led Program for Parents of Extremely Pre-term Infants
Brief Title: Therapist Education and Massage for Parent Infant-Outcomes
Acronym: TEMPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-0282; KL2TR002490 (NIH)
Record Dates: First submitted 2019-10-04; First posted 2019-10-10 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Parent-Child Relations; Parents; Extreme Prematurity
MeSH Terms: interventions — Massage

STUDY DESIGN:
Intervention Model Description: Prospective single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEMPO (Experimental): The Therapist Education and Massage for Parent-Infant Outcomes program (TEMPO) is a structured, therapist-led physical therapy program. TEMPO trains and supports parents to deliver physical therapy interventions including massage and developmental play during hospitalization and in the home setting.
  Interventions: Other: Therapist Education and Massage for Parents of Extremely Preterm Infants

INTERVENTIONS:
Other: Therapist Education and Massage for Parents of Extremely Preterm Infants — TEMPO includes these components:
  * Early Parent Education Session
  * Weekly Parent Education Sessions
  * Infant Massage Parent Education Sessions
  * Discharge Parent Education Session
  * Parent Education Post-Discharge
  * Bi-weekly emails (or texts)
  * 2 Month Follow-up Massage Review Session

SUMMARY:
The Therapist Education and Massage for Parent-Infant Outcomes program is evidence-based and includes infant massage, physical therapy interventions including developmental support and play activities to promote infant behavioral-motor development, principles of family-centered care, and multiple modes of educational delivery to enhance parent retention of knowledge, parent-infant bonding, and confidence in continuing physical therapy interventions after discharge.

DETAILED DESCRIPTION:
The Therapist Education and Massage for Parent-Infant Outcomes program involves components during and after hospitalization.

During infant hospitalization • Visit 1: Early Parent Education Session: Initiated within 3 weeks of infant birth. The therapist will educate the parent about the importance of infant positioning, the impact of prematurity on the motor and sensory systems, and how to read and respond to infant behavioral-motor cues using a written pamphlet with pictures to supplement the verbal education lasting about 30 minutes.

* The therapist will ask the parent to complete a contact information form and a demographic form and a baseline questionnaire.

  * Visits 2-8: Weekly Parent Education Sessions <34 weeks: Following the initial parent education session, the therapist will hold weekly parent education sessions, ideally at the time of therapy. When the infant is this young (<34 weeks gestation), therapist intervention and education will focus on infant behavioral-motor cues, reading/response to infant cues, positioning strategies/concerns, and developmentally appropriate stimulation of the infant. If the parent is not available for all therapy sessions, then the parent will receive a weekly update about their infant's progress face-to-face and/or via video chat.
  * Visits 9-10: Infant Massage Parent Education Sessions: Parent-administered infant massage will be incorporated into the therapy plan of care as soon as the infant's medical provider determines that the infant is physiologically stable and can tolerate massage. This time is generally once the infant is approximately 34 weeks gestational age, approximately 1500 grams, and is demonstrating temperature stability out of the isolette for short periods. At a minimum, the therapist will teach massage for the back or lower extremities over 2 parent education sessions. The therapist will demonstrate massage strokes on a doll using verbal cues to guide the parent while the parent administers massage on the infant. An instructional massage pamphlet will be provided. Once the therapist has determined parent safety with massage administration, parents will be encouraged to practice infant massage when they visit the baby and to note when they do this by marking a card at the bedside.
* Pre and Post both massage sessions, the Primary Investigator or study coordinator will collect salivary cortisol via buccal swab as a measure of physiologic stress.

  * Visits 11+: Weekly Parent Education Sessions >34 weeks: Weekly parent education once the infant is >34 weeks will begin to incorporate hands-on developmental play activities, introduction to visual engagement, and postural control practice in variety of positions that the infant tolerates. Additionally, the therapist and parent may choose to review massage at these visits. If the parent is not available for all therapy sessions, then the parent will receive a weekly update about their infant's progress face-to-face and/or via video chat.
  * Final Visit during hospitalization: Within the week of hospital discharge, the therapist will schedule a face-to-face parent education session lasting about 30 minutes to review age-appropriate developmental play activities for home and review infant massage. A supplemental handout and therapist email and pager information will be provided.
* At this visit, the therapist will have the parent fill out a questionnaire.

Follow- up procedures (by visits) The program has additional components that extend beyond the hospital period. Parent and infant outcome measures will be collected at the first follow-up and 12 month corrected age follow-up clinic visits.

After hospitalization:

* Visit 1: Parent Education Post-Discharge: The therapist will call the parent within 2 weeks of discharge to follow up about discharge education and massage. During this phone call, the therapist will review the home program and massage techniques. The therapist will also answer any parent questions. Therapist email and pager information will be provided.
* Visits 2-12 (approximate): Bi-weekly emails (or texts): The therapist will send bi-weekly emails or texts (depending on parents' preference) with developmental play activity and massage reminders and tips from hospital discharge through the first follow up appointment.
* Visit 13 (approximate): First Visit Follow-up Massage Review Session: At the infant's first follow-up appointment with the multidisciplinary neonatology team, the therapist will provide a gross motor screening assessment and education. In addition, as part of the program, a therapist will facilitate a parent-administered infant massage session to provide an opportunity for parent to receive feedback on technique from the therapist. This session will address any safety concerns, infant changes, and parent questions.

  o At this visit, the therapist will have the parent fill out a questionnaire for ongoing measurement.
* Visits 14+ (approximate): Bi-weekly emails (or texts): The therapist will continue to send bi-weekly emails or texts (depending on parents' preference) with developmental play activity and massage reminders until the 12 month followup appointment.
* 12 Month Follow-up Appointment: At the standard of care 12 month corrected age follow-up appointment with the multidisciplinary neonatology team, the PI or study coordinator will interview the parent about acceptability of the program.

  * At this visit, the therapist will have the parent fill out a questionnaire for ongoing measurement

ELIGIBILITY:
Inclusion Criteria:

* Infants with gestational age <28 weeks gestation, within the first 3 weeks of life, and their
* Biologic mother or father must be able to speak and understand English.

Exclusion Criteria:

* Infants who do not have a biological parent available to consent within the first 3 weeks of life.
* Infants with genetic/chromosomal abnormality, congenital neurological or musculoskeletal disorder, or abnormal bone density related to a congenital condition that would affect the ability to do massage and/or exercise and the safety of the infant.
* Parents who are unwilling to engage in all components of TEMPO.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana McCarty, DPT, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Children's Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the university.
Supporting Information: CSR
Time Frame: NIH expects the timely release and sharing of data to be no later than the acceptance for publication of the main findings from the final dataset. Publication is anticipated within one year of the study conclusion.
Access Criteria: Data use agreement. http://research.unc.edu/clinical-trials/clinical-trials-gov/data-sharing-guidance/
URL: http://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm

REFERENCES:
- See also: NIH Data Sharing Policy — http://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- TEMPO: The Therapist Education and Massage for Parent-Infant Outcomes program (TEMPO) is a structured, therapist-led physical therapy program. TEMPO trains and supports parents to deliver physical therapy interventions including massage and developmental play during hospitalization and in the home setting.
  Therapist Education and Massage for Parents of Extremely Preterm Infants: TEMPO includes these components:
  * Early Parent Education Session
  * Weekly Parent Education Sessions
  * Infant Massage Parent Education Sessions
  * Discharge Parent Education Session
  * Parent Education Post-Discharge
  * Bi-weekly emails (or texts)
  * 2 Month Follow-up Massage Review Session
Period: Overall Study
Arm/Group | TEMPO
Started | 68
Parents | 32
Infants | 36
Completed | 37
Not Completed | 31

BASELINE CHARACTERISTICS:
Groups:
- TEMPO Parents: The Therapist Education and Massage for Parent-Infant Outcomes program (TEMPO) is a structured, therapist-led physical therapy program. TEMPO trains and supports parents to deliver physical therapy interventions including massage and developmental play during hospitalization and in the home setting.
  Therapist Education and Massage for Parents of Extremely Preterm Infants: TEMPO includes these components:
  * Early Parent Education Session
  * Weekly Parent Education Sessions
  * Infant Massage Parent Education Sessions
  * Discharge Parent Education Session
  * Parent Education Post-Discharge
  * Bi-weekly emails (or texts)
  * 2 Month Follow-up Massage Review Session
- TEMPO Infants: Physical Therapy (PT) and Occupational Therapy (OT) Initial Assessment: Initiated within the first 72-96 hours of life (if infant medically stable)
  * PT and OT Intervention at <33 weeks Post Menstrual Age (PMA): During hospitalization, infants received PT and OT intervention 4-5 times weekly (total) for approximately 15-30 minutes at a time.
  * PT and OT Re-assessment: Performed between 33-34 weeks PMA if infant was physiologically stable.
  * PT and OT Intervention >33 weeks PMA: Infants continued to receive combined PT or OT intervention 4-5 times weekly for approximately 30 minutes.
  * Discharge Education: In standard of care therapy, the PT or OT reviewed a 2-page handout with the parent if they are available at the bedside the week of discharge.
  * <4 month and 12-month Follow-Up Visits: The Special Infant Care Clinic is a multidisciplinary follow-up clinic that follows the neurodevelopment of preterm infants discharged from the Neonatal Critical Care Center (NCCC).
- Total: Total of all reporting groups
Arm/Group | TEMPO Parents | TEMPO Infants | Total
Number analyzed (Participants) | 32 | 36 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 36 | 36
  Between 18 and 65 years | 32 | 0 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 20 | 51
  Male | 1 | 16 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 28 | 32 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 17 | 20 | 37
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 7 | 7 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 36 | 68

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eligible Dyads Who Would Consent to Enroll (Recruitment)
Description: Recruitment is defined as the percent of eligible participants enrolled of those approached.
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 35
percentage of participants | 91

2. Primary Outcome: Percent of Parents Who Would Recommend This Program to Other Parents of Preterm Infants
Description: The percent of enrolled parents who report they would recommend the program to other parents.
Time Frame: Final follow up visit - an average of 15-18 months after study period begins
Population: Includes all parents who were retained through the final Follow Up visit.
Measure: Number; unit: percentage of participants
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 18
percentage of participants | 100

3. Primary Outcome: Percent of Parents Who Complete All Protocol Components (Adherence)
Description: The percent of enrolled parents who complete all protocol components during hospitalization.
Time Frame: At hospital discharge, approximately 8-16 weeks after enrollment
Population: Six parents transferred to an outside hospital and 3 infants died prior to hospital discharge; therefore, 23 dyads were maintained at hospital discharge.
Measure: Number; unit: percentage of participants
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 23
percentage of participants | 87

4. Primary Outcome: Percent of Parents Who Are Retained in the Study at 12 Months (Retention)
Description: Percent of enrolled parents who are retained in the study at 12 months.
Time Frame: Final follow up visit - an average of 15-18 months after study period begins
Population: More parents agreed to a phone interview than those who agreed to return their child for testing.
Measure: Number; unit: percentage of participants
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 32
percentage of participants | 56

5. Primary Outcome: Percent of Enrolled Parents Who Provide Complete Data and Interviews
Description: The percent of enrolled parents who provide complete data and interviews.
Time Frame: Final follow up visit - an average of 15-18 months after study period begins
Measure: Number; unit: percentage of participants
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 32
percentage of participants | 56

6. Primary Outcome: Average Number of Days Per Week That Enrolled Parents Complete TEMPO Activities
Description: The average days per week that parents completed TEMPO activities based on parents' weekly self reports.
Time Frame: at First follow up visit - approximately 1 to 2 months after hospital discharge
Population: Includes number of parents interviewed at first Follow up visit.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 17
days per week | 4.5 (1.5)

7. Primary Outcome: Percent of Parents Who Rate Acceptability as 4/5 or 5/5 Using the Acceptability of Intervention Measure
Description: Longitudinal measures of parents' perceived acceptability of intervention throughout the study period measured by the percent of parents who rate acceptability as 4/5 or 5/5 using the Acceptability of Intervention Measure. The Acceptability of Intervention Measure is a 12 item implementation outcome assessment designed to measure if the intervention is perceived as agreeable, palatable, or satisfactory. Cut-off scores for interpretation are not yet available; however, higher scores indicate greater acceptability.
Time Frame: Baseline, Hospital Discharge (Variable 8-12 weeks), First Follow up (at 1-2 months post discharge), Second Follow up (at 15-18 months)
Population: Data reported for all parents who responded to surveys at the specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 32
percentage of participants
  Baseline | 81
  Hospital Discharge: number analyzed (Participants) | 23
  Hospital Discharge | 95
  First Follow Up: number analyzed (Participants) | 10
  First Follow Up | 100
  Second Follow Up: number analyzed (Participants) | 12
  Second Follow Up | 91

8. Primary Outcome: Percent of Parents Who Rate Acceptability as 4/5 or 5/5 Using the Feasibility of Intervention Measure
Description: Longitudinal measures of parents' perceived feasibility of intervention throughout the study period measured by the percent of parents who rate feasibility as 4/5 or 5/5 using the Feasibility of Intervention Measure. The Feasibility of Intervention Measure is a 9 item implementation outcome assessment designed to measure the extent to which a new treatment can be successfully used or carried out. Cut-off scores for interpretation are not yet available; however, higher scores indicate greater feasibility.
Time Frame: as for outcome 7
Population: Data reported for all parents who responded to surveys at the specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 32
percentage of participants
  Baseline | 78
  Hospital Discharge: number analyzed (Participants) | 23
  Hospital Discharge | 100
  First Follow Up: number analyzed (Participants) | 10
  First Follow Up | 100
  Second Follow Up: number analyzed (Participants) | 12
  Second Follow Up | 91

9. Primary Outcome: Qualitative Summaries of Parent Experience Via Interview
Description: The Primary Investigator or research coordinator will conduct interviews with parents at both follow up visits using 3 questions developed by the Primary Investigator to assess feasibility, acceptability, and perceived benefit of massage. Yes/No responses were provided for the following questions: (1) "Was it difficult to meet the therapist weekly for TEMPO sessions?"; (2) "Would you recommend TEMPO to other parents of preterm infants?"; and (3) "Have you continued doing massage with your baby at home?".
Time Frame: First follow up visit - an average of 6-10 months after study period begins; Final follow up visit - an average of 15-18 months after study period begins
Population: Responses reported for participants who answered "yes".
Measure: Number; unit: percentage of participants
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 19
percentage of participants
  Feasibility | 95
  Acceptability | 100
  Perceived benefit | 95

10. Secondary Outcome: Mean Infant Salivary Cortisol Level
Description: Buccal swab will be taken immediately pre and post massage implementation during hospitalization at the massage education session with therapist. Sample means and standard deviations will be reported to provide an estimate of population parameters needed for planning a future study. Salivary cortisol is a biomarker for stress15 that may be used to understand the mechanism by which the intervention impacts physiological stress states.
Time Frame: To be measured twice immediately pre-and post initial massage education in the hospital.
Population: Both a pre- and post initial massage sample was required to detect & report change and no sufficient samples were collected for any infant at both timepoints. Insufficient (or immeasurable) samples were collected for all infants across all timepoints.
Groups:
- TEMPO Infants: PT and OT Initial Assessment: Initiated within the first 72-96 hours of life (if infant medically stable)
  * PT and OT Intervention at <33 weeks PMA: During hospitalization, infants received PT and OT intervention 4-5 times weekly (total) for approximately 15-30 minutes at a time.
  * PT and OT Re-assessment: Performed between 33-34 weeks PMA if infant was physiologically stable.
  * PT and OT Intervention >33 weeks PMA: Infants continued to receive combined PT or OT intervention 4-5 times weekly for approximately 30 minutes.
  * Discharge Education: In standard of care therapy, the PT or OT reviewed a 2-page handout with the parent if they are available at the bedside the week of discharge.
  * <4 month and 12-month Follow-Up Visits: The Special Infant Care Clinic is a multidisciplinary follow-up clinic that follows the neurodevelopment of preterm infants discharged from the NCCC.
Arm/Group | TEMPO Infants
Number analyzed (Participants) | 0

11. Secondary Outcome: Parent Salivary Cortisol Level
Description: Sample means and standard deviations will be reported to provide an estimate of population parameters needed for planning a future study. Salivary cortisol is a biomarker for stress 15 that may be used to understand the mechanism by which the intervention impacts physiological stress states. Paired t-tests were conducted to assess pre- to post-infant massage cortisol levels in parents.
Time Frame: To be measured twice immediately pre-and post initial massage education in the hospital. Buccal swab will be taken immediately pre and post massage implementation during hospitalization at the massage education session with therapist.
Population: Six parents transferred to an outside hospital and 3 infants died prior to hospital discharge; therefore, 23 dyads were maintained at hospital discharge. One additional male parent was excluded from analysis because salivary cortisol is sex-specific.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 22
ng/dL | -18.05 (34.89)
Statistical Analysis 1: Comparison: TEMPO Parents; Test type: Other; p = 0.024, t-test, 2 sided

12. Secondary Outcome: Bayley Scales of Infant Development IV
Description: The Bayley Scales of Infant Development IV (BSID-IV) is a standardized assessment to evaluate cognitive development, expressive and receptive language, and fine and gross motor development in children between the ages of 1 and 42 months. For the purpose of this study, only the gross motor scale was recorded. For infants at approximately 12 months corrected, the total gross motor scaled scores range from 0-19 with 0 indicating the highest risk of developmental delay and 19 indicating the lowest risk of developmental delay.
Time Frame: Final follow up visit - an average of 15-18 months after study period begins
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | TEMPO Infants
Number analyzed (Participants) | 11
score on a scale | 11.6 [7 to 13]

13. Secondary Outcome: Longitudinal Measures in Patient-Reported Outcomes Measurement Information System Adult Profile Short Form - Anxiety
Description: Sample medians and standard deviations will be reported to provide an estimate of population parameters needed for planning a future study. An 8 item validated measure with each item rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of anxiety.
Time Frame: as for outcome 7
Population: Although 32 parents were enrolled, Baseline survey data was only collected for 24 . Hospital discharge data was collected for 19 parents. All data were reported for parents who were not lost to follow up.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 24
score on a scale
  Baseline | 20 (5.28)
  Hospital Discharge: number analyzed (Participants) | 19
  Hospital Discharge | 12 (4.03)
  First Follow Up: number analyzed (Participants) | 9
  First Follow Up | 10 (5.27)
  Second Follow Up: number analyzed (Participants) | 12
  Second Follow Up | 9.5 (3.61)

14. Secondary Outcome: Longitudinal Measures in Centers for Epidemiologic Studies Depression Scale
Description: Sample means and standard deviations will be reported to provide an estimate of population parameters needed for planning a future study. A valid, reliable self-assessment tool for evaluating depressive symptoms in adult populations, including among mothers during and after parturition. The 20 item form will be used. Possible range of scores is 0-60, with the higher scores indicating the presence of more symptomatology.
Time Frame: as for outcome 7
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 24
score on a scale
  Baseline | 15.4 (7.59)
  Hospital Discharge: number analyzed (Participants) | 19
  Hospital Discharge | 8.21 (4.85)
  First Follow Up: number analyzed (Participants) | 9
  First Follow Up | 8.0 (3.84)
  Second Follow Up: number analyzed (Participants) | 12
  Second Follow Up | 7.83 (5.46)

15. Secondary Outcome: Longitudinal Measures Changes in Edinburgh Postnatal Depression Scale
Description: Sample means and standard deviations will be reported to provide an estimate of population parameters needed for planning a future study. A 10-item self-report questionnaire validated to detect change in depressive symptoms in mothers both during and after the postnatal period. Scores range from 0-30, with scores greater than 13 indicating likely depressive illness.
Time Frame: as for outcome 7
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 24
score on a scale
  Baseline | 17.2 (2.19)
  Hospital Discharge: number analyzed (Participants) | 19
  Hospital Discharge | 18.36 (2.10)
  First Follow Up: number analyzed (Participants) | 9
  First Follow Up | 18.7 (2.18)
  Second Follow Up: number analyzed (Participants) | 12
  Second Follow Up | 19.2 (2.18)

16. Secondary Outcome: Longitudinal Measures Changes in Parenting Sense of Competence Scale
Description: Sample means and standard deviations will be reported to provide an estimate of population parameters needed for planning a future study. A 17-item scale using ratings (Strongly Disagree-1, Somewhat Disagree-2, Disagree-3, Agree-4, Somewhat Agree-5, Strongly Agree-6) to assess satisfaction of parenting and parental self-efficacy in a variety of populations with a range in score from 17 to 102 and higher scores indicating a greater sense of parental self-efficacy.
Time Frame: as for outcome 7
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TEMPO Infants
Number analyzed (Participants) | 24
score on a scale
  Baseline | 76.6 (9.99)
  Hospital Discharge: number analyzed (Participants) | 19
  Hospital Discharge | 82.61 (9.88)
  First Follow Up: number analyzed (Participants) | 9
  First Follow Up | 85.0 (11.88)
  Second Follow Up: number analyzed (Participants) | 12
  Second Follow Up | 87.2 (10.71)

17. Secondary Outcome: Postnatal Attachment Questionnaire
Description: Sample means and standard deviations will be reported to provide an estimate of population parameters needed for planning a future study. A Maternal Postnatal Attachment Scale (MPAS) with 19 items representing 4 components: pleasure in proximity, tolerance, need-gratification and protection, and knowledge acquisition was used to query the parents' feelings about their infants under 1 year of age. The MPAS is a self-reported scale to reflect the degree of subjective emotional connection between mothers and their infants.The scale includes two, three, four and five options.The total score span of the scale is between 19-95, and the higher the score, the higher the level of maternal and child attachment.
Time Frame: Final follow up visit - an average of 15-18 months after study period begins
Population: All data were reported for parents who were not lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 12
score on a scale | 87.9 (5.9)

18. Secondary Outcome: Longitudinal Measures in Infant Temperament Using Carey Temperament Scales
Description: Sample means and standard deviations will be reported to provide an estimate of population parameters needed for planning a future study. This questionnaire assesses nine temperamental characteristics of infants. Caregivers are presented with a statement describing a certain behavior and asked to rate how often their child behaves in that way on a scale from 1 (almost never) to 6 (almost always), with higher scores indicating more difficult temperament
Time Frame: as for outcome 9
Population: In order to limit parent burden, the investigators removed this questionnaire from the survey battery.
Arm/Group | TEMPO Parents
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for infants only from the time of parental informed consent through hospital discharge, approximately 8-16 weeks after enrollment. Since infants were the only population considered to be as risk, adverse events were not collected for parents.
Groups:
- TEMPO Infants: PT and OT Initial Assessment: Initiated within the first 72-96 hours of life (if infant medically stable) PT and OT Intervention at <33 weeks PMA: During hospitalization, infants received PT and OT intervention 4-5 times weekly (total) for approximately 15-30 minutes at a time.
  PT and OT Re-assessment: Performed between 33-34 weeks PMA if infant was physiologically stable.
  PT and OT Intervention >33 weeks PMA: Infants continued to receive combined PT or OT intervention 4-5 times weekly for approximately 30 minutes.
  Discharge Education: In standard of care therapy, the PT or OT reviewed a 2-page handout with the parent if they are available at the bedside the week of discharge.
  <4 month and 12-month Follow-Up Visits: The Special Infant Care Clinic is a multidisciplinary follow-up clinic that follows the neurodevelopment of preterm infants discharged from the NCCC.
Arm/Group | TEMPO Infants
All-Cause Mortality (participants affected / at risk) | 3/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT04121897/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT04121897/ICF_001.pdf